CLINICAL TRIAL: NCT05144139
Title: A Phase I/II Clinical Trial to Evaluate the Safety, Immunogenicity and Immune Persistence of COVID-19 mRNA Vaccine in Healthy People Aged 18 Years and Above.
Brief Title: A Phase I/II Clinical Trial in Healthy People Aged 18 Years and Above
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stemirna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: SWC002
Record Dates: First submitted 2021-11-11; First posted 2021-12-03 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-10

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19 | interventions — CVnCoV COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low dose group with mRNA vaccine (Experimental): 25μg with COVID-19 mRNA vaccine
  Interventions: Biological: COVID-19 mRNA vaccine
- Low dose group with placebo (Placebo Comparator): Low dose group with placebo
  Interventions: Biological: COVID-19 mRNA vaccine
- High dose group with mRNA vaccine (Experimental): 45μg with COVID-19 mRNA vaccine
  Interventions: Biological: COVID-19 mRNA vaccine
- High dose group with placebo (Placebo Comparator): High dose group with placebo
  Interventions: Biological: COVID-19 mRNA vaccine

INTERVENTIONS:
Biological: COVID-19 mRNA vaccine — Intramuscular injection, COVID-19 mRNA vaccine/placebo, 21 days interval

SUMMARY:
This clinical trial is a phase I/II clinical trial to evaluate the safety, immunogenicity and immune persistence of COVID-19 mRNA vaccine in healthy people aged 18 years and above.

DETAILED DESCRIPTION:
This is the clinical trial including an open-label, single-arm Phase I study and a subsequent randomized, blind, placebo-parallel controlled Phase II study to evaluate the safety, immunogenicity and immune persistence of COVID-19 mRNA vaccine in healthy people aged 18-60 years and ≥18 years respectively, whose locations or circumstances put them at appreciable risk of acquiring COVID-19 and/or SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* People aged 18-60 years (both inclusive) for phase 1 and aged ≥18 years for phase 2；
* Medical history and physical examination indicating as a healthy person;
* The female participant or the spouse (or partner) of the male participant in child-birthing age agrees to use effective contraceptive measure throughout the whole course of this clinical trial.
* Those who are participating in this clinical trial voluntarily, have signed the informed consent form, and been able to understand and comply with the requirements of the clinical trial protocol.

Exclusion Criteria:

* Confirmed cases or history of SARS-CoV-2 infection;
* Has a history of SARS and MERS virus infection;
* Has fever (axillary temperature ≥37.3℃), dry cough, fatigue, nasal congestion, runny nose, sore throat, myalgia, diarrhea, shortness of breath, and dyspnea within 14 days before vaccination;
* Positive urine pregnancy test；
* Axillary temperature ≥37.3℃ at the day vaccinated;
* History of severe allergic reactions to vaccination (such as acute allergic reactions, urticaria, dyspnea, angioneurosis, edema, etc.) or allergies to known components of COVID-19 mRNA vaccine;
* History or family history of convulsions, epilepsy, encephalopathy, or mental illness;
* Suffering from congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.;
* Known suffering from diseases including: acute respiratory disease (such as flu-like illness, acute cough, sore throat), severe cardiovascular disease, kidney disease, uncontrolled hypertension (systolic blood pressure >150 mmHg, diastolic blood pressure >90 mmHg), diabetes complications, malignant tumor, all sorts of acute illness or chronic diseases acute phase;
* Diagnosis with congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, or other autoimmune disease;
* Abnormal coagulation function (such as lack of coagulation factor, coagulation disorders);
* Receiving anti-tuberculosis treatment;
* Long-term receipt (continuous≥7 days) of glucocorticoid (reverence value for dose: amount to≥20 mg/d prednisone equivalent), except inhaled, topical, nasal, aural and ophthalmic corticosteroids, within 6 months before screening; Receipt of immunotherapy or immunosuppressant within 3 months (continuous oral or infusion for more than 14 days);
* Receipt of live attenuated vaccine within 28 days prior to vaccination and other vaccines within 14 days prior to vaccination;
* Receipt of blood products within 3 months prior to vaccination
* Receipt of other study drugs within 6 months prior to vaccination;
* Receipt of any SARS-COV-2 vaccine;
* Other situations judged by the investigators that are not suitable for participating in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2022-08-28 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
local/systemic solicited adverse reaction/events | up to 6 days after each dose
  The incidence of local/systemic solicited adverse reaction/events
unsolicited adverse events | up to 21 days and up to 28 days after the first and second dose of immunization, respectively
  The incidence of unsolicited adverse events
The incidence of SAE | up to 28 days after the full course of immunization
  The incidence of SAE from the first dose of vaccination to 28 days after the full course of immunization

SECONDARY OUTCOMES:
The seroconversion rate, 2-fold or 4-fold rise and GMT/GMI of the SARS-COV-2 S-protein specific antibody (specific total antibody/IgG antibody) and neutralizing antibody | 14 days after the full immunization
  The seroconversion rate, 2-fold or 4-fold rise and GMT/GMI of the SARS-COV-2 S-protein specific antibody (specific total antibody/IgG antibody) and neutralizing antibody 14 days after the full immunization in the subjects who take two doses as protocol specified
The incidence of SAE | the 29th ~365th day after the full course of immunization
  The incidence of SAE within the 29th ~365th day after the full course of immunization
Changes in laboratory abnormal parameters | after at least of one dose
  Changes in laboratory abnormal parameters in the participants who take at least of one dose

OTHER OUTCOMES:
The positive conversion rate, 2-fold or 4-fold rise and GMT/GMI of the SARS-COV-2 S-protein specific antibody (specific total antibody/IgG antibody), neutralizing antibody | before 1st and 2nd immunization, 90, 180, 365 days after the full immunization
  The positive conversion rate, 2-fold or 4-fold rise and GMT/GMI of the SARS-COV-2 S-protein specific antibody (specific total antibody/IgG antibody), neutralizing antibody before 1st and 2nd immunization, 90, 180, 365 days after the full immunization
Cellular immunity INF-γ, IL-4 and IL-2 | before 1st and 2nd immunization, and 14, 90, 180, 365 days after the full immunization
  Cellular immunity (INF-γ, IL-4 and IL-2) before 1st and 2nd immunization, and 14, 90, 180, 365 days after the full immunization

CONTACTS AND LOCATIONS:
Overall Officials: Mayfong Mayxay, professor, Principal Investigator — Mahosot Hospital
Locations (1):
- Mayfong Mayxay, Vientiane, Laos

IPD SHARING:
Plan to Share IPD: No